CLINICAL TRIAL: NCT00456807
Title: Complementary Testing to Further Evaluate the Immunogenicity of a GSK Biologicals' HPV Vaccine (580299) in Healthy Female Subjects Aged Over 26 Years Enrolled in Study 104820.
Brief Title: Complementary Testing to Evaluate Immunogenicity of Human Papillomavirus (HPV) Vaccine (580299) in Healthy Female Subjects Aged >/= 26 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 109801
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Results first posted 2010-07-30 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: Human Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cervarix Group (Experimental): Subjects who received 3 doses of Cervarix during the primary study (NCT00294047).
  Interventions: Biological: Cervarix TM
- Placebo Group (Placebo Comparator): Subjects who received 3 doses of placebo during the primary study (NCT00294047).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Placebo Group
Biological: Cervarix TM — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Other Names: GSK Biologicals' HPV-16/18 VLP/AS04 vaccine
  Arms: Cervarix Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. Indeed, certain oncogenic types of HPV can infect the cervix (part of the uterus or womb). This infection may go away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. This study will supplement an ongoing study evaluating the safety, efficacy and immunogenicity of the vaccine in women aged 26 years and above. This study will therefore assess additional immunogenicity parameters of the vaccine in women from selected investigative sites.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* A female enrolled in study 104820 and who received three doses of study vaccine/control.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the subject prior to enrolment in this ancillary study.

Exclusion Criteria:

* Pregnancy.
* Administration of any HPV vaccine other than that foreseen by the study protocol.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine since study start.
* Chronic administration of immunosuppressants or other immune-modifying drugs since study start.
* Administration of immunoglobulins and/or any blood products within 90 days preceding a blood sampling.

Min Age: 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Netherlands (2):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Delft

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109801 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at pre-selected sites in the primary study HPV-015 (NCT00294047) who were in the immunogenicity subset and have received all three doses of vaccine/control were asked to participate in the present ancillary study.
Pre-assignment Details: This ancillary study will consist of supplemental testing of serological and cervical samples obtained at Visit 5 (Month 12) and Visit 6 (Month 18) of the primary study HPV-015 (NCT00294047) from pre-selected sites.
Period: Overall Study
Arm/Group | Cervarix Group | Placebo Group
Started | 53 | 47
Completed | 52 | 47
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 53 | 47 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (8.44) | 40.3 (8.83) | 40.6 (8.63)
Gender [Count of Participants; unit: Participants]
  Female | 53 | 47 | 100
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Cytokine-positive CD4/CD8 Cells Per Million in Tests Producing at Least 2 Different Cytokines
Description: The geometric mean and 95% confidence interval of the number of Human Papilloma Virus type 16 (HPV-16) and HPV-18 specific CD4 and CD8 cells producing at least 2 different cytokines is reported per million of CD4 or CD8 T-cells, respectively.
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on subjects from the Total Vaccinated Cohort with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: cells per million CD4/CD8 T-cells
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 52 | 47
cells per million CD4/CD8 T-cells
  HPV-16 specific CD4 [Month 12] (n=52,46) | 877.4 [665.0 to 1157.7] | 19.5 [9.4 to 40.5]
  HPV-16 specific CD4 [Month 18] (n=52,47) | 738.5 [512.9 to 1063.3] | 22.3 [11.3 to 44.0]
  HPV-16 specific CD8 [Month 12] (n=52,46) | 2.0 [1.3 to 3.1] | 2.0 [1.2 to 3.1]
  HPV-16 specific CD8 [Month 18] (n=50,47) | 2.9 [1.8 to 4.7] | 2.7 [1.6 to 4.6]
  HPV-18 specific CD4 [Month 12] (n=52,46) | 581.2 [428.0 to 789.2] | 11.5 [5.7 to 23.4]
  HPV-18 specific CD4 [Month 18] (n=52,47) | 300.1 [171.9 to 524.1] | 16.8 [9.1 to 31.2]
  HPV-18 specific CD8 [Month 12] (n=52,46) | 2.1 [1.3 to 3.3] | 1.8 [1.1 to 2.7]
  HPV-18 specific CD8 [Month 18] (n=50,47) | 2.8 [1.7 to 4.6] | 4.7 [2.6 to 8.7]

2. Primary Outcome: Number of B-cells Per Million Showing a Specific Memory Response for HPV-16 and HPV-18
Description: The geometric mean and 95% confidence interval of the number of HPV-16 and HPV-18 specific memory B-cells is reported per million of B-cells.
  An arbitrary value of 0 was given for subjects with antibody concentration below the limit of quantification.
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on subjects from the Total Vaccinated Cohort with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: cells per million B-cells
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 51 | 45
cells per million B-cells
  HPV-16 specific [Month 12] (n=51,44) | 517.1 [361.4 to 739.9] | 101.4 [45.1 to 227.9]
  HPV-16 specific [Month 18] (n=51,45) | 304.4 [210.0 to 441.1] | 33.1 [6.7 to 163.0]
  HPV-18 specific [Month 12] (n=51,44) | 354.7 [253.1 to 497.1] | 68.4 [27.0 to 173.2]
  HPV-18 specific [Month 18] (n=51,45) | 301.5 [223.9 to 406.0] | 0.0 [0 to 0]

3. Primary Outcome: Number of Subjects With Anti-HPV-16 and Anti-HPV-18 Antibody Concentrations Above Pre-defined Cut-off Values
Description: Cut-off values assessed include 8 enzyme-linked immunosorbent assay units Per Milliliter (EL.U/mL)for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on subjects from the Total Vaccinated Cohort with available results.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 52 | 46
Subjects
  Anti-HPV-16 [Month 12] (n=52, 45) | 52 | 14
  Anti-HPV-16 [Month 18] (n=49, 46) | 49 | 14
  Anti-HPV-18 [Month 12] (n=52, 45) | 52 | 7
  Anti-HPV-18 [Month 18] (n=49, 46) | 49 | 7

4. Primary Outcome: Titers of Anti-HPV-16 and Anti-HPV-18 Antibodies
Description: Titers are presented as Geometric Mean Titers (GMTs).
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on subjects from the Total Vaccinated Cohort with available results.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 52 | 46
Titer
  Anti-HPV-16 [Month 12] (n=52, 45) | 2050.4 [1456.1 to 2887.3] | 6.9 [5.3 to 9.0]
  Anti-HPV-16 [Month 18] (n=49, 46) | 1517.1 [1067.4 to 2156.4] | 7.2 [5.4 to 9.5]
  Anti-HPV-18 [Month 12] (n=52, 45) | 761.4 [538.0 to 1077.5] | 4.8 [3.5 to 6.7]
  Anti-HPV-18 [Month 18] (n=49, 46) | 551.4 [387.5 to 784.6] | 4.9 [3.6 to 6.6]

5. Primary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) Immunoglobulin G (IgG) Antibodies
Description: Titers given as Geometric Mean Titers (GMTs). An arbitrary value of 0 was given for subjects with antibody concentration below the limit of quantification.
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data. None of the subjects in the Placebo Group had detectable antibodies against HPV-16 at Months 12 and 18 and against HPV-18 at Month 12.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 26 | 20
Titer
  Anti-HPV16 [Month 12] (n=12, 10) | 129.5 [58.0 to 289.2] | 0 [0 to 0]
  Anti-HPV16 [Month 18] (n=26, 20) | 99.9 [48.9 to 203.8] | 0 [0 to 0]
  Anti-HPV18 [Month 12] (n=12, 10) | 67.2 [28.6 to 158.0] | 0 [0 to 0]
  Anti-HPV18 [Month 18] (n=26, 20) | 42.8 [23.1 to 79.6] | 5.8 [5.8 to 5.8]

6. Primary Outcome: Correlation of Anti-HPV-16 and Anti-HPV-18 Antibodies in Serum and in Cervical Secretion (CVS) Samples
Description: Pearson coefficients of correlation between serum and CVS for anti-HPV-16 and anti-HPV-18 titers standardized for total IgG were calculated.
Time Frame: At Month 12 and Month 18 after first vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, only on those subjects from the Cervarix group with CVS sample results available.
Measure: Number; unit: correlation coefficient
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 26 | 0
correlation coefficient
  Anti-HVP-16 (Month 12) | 0.903 |
  Anti- HPV-16 (Month 18) | 0.898 |
  Anti-HPV-18 (Month 12) | 0.901 |
  Anti-HPV-18 (Month 18) | 0.876 |

ADVERSE EVENTS:
Description: No safety data were collected in the framework of this ancillary study.
Arm/Group | Cervarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No safety data were collected in the framework of this ancillary study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.